CLINICAL TRIAL: NCT05682703
Title: A Bidirectional Study in Exploring the Dynamic Changes of Plasma and Urine Metabolites During the Occurrence and Development of Nasopharyngeal Carcinoma in Southern China.
Brief Title: A Bidirectional Study in Exploring the Dynamic Changes of Plasma and Urine Metabolites of Nasopharyngeal Carcinoma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-470
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Nasopharyngeal Carcinoma; EBV Infection
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Plasma and Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EBV virus infector: QPCR/EBV antibody, diagnosed as EBV infection patient
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy
- nasopharyngeal carcinoma patients: Patients diagnosed as nasopharyngeal carcinoma by pathological diagnosis (2018 WHO standard)
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy
- Healthy people: healthy people with no history of nasopharynx related diseases or other known diseases that may affect blood lipid/protein metabolism
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy

INTERVENTIONS:
Diagnostic Test: Proteomics technology and liquid biopsy — using proteomics technology and liquid biopsy to investigate the changes of plasma and urine metabolites by collecting residual blood and urine from routine diagnosis and treatment or physical examination

SUMMARY:
The transformation process of nasopharyngeal carcinoma is complex, so it is particularly important to explore the relationship between various disease states on its clinical pathway. Therefore, we carried out this study to explore the changes of plasma and urine metabolites at different stages during the occurrence and development of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* EBV virus infector: QPCR/EBV antibody, diagnosed as EBV infection patient with previous infection;
* Nasopharyngeal carcinoma patients:Patients diagnosed as nasopharyngeal carcinoma by pathological diagnosis (2018 WHO standard);
* Healthy people: Healthy people who have no history of nasopharynx related diseases or other known diseases that may affect blood lipid/protein metabolism and have been hospitalized in the Physical Examination Center of Southern Hospital.

Exclusion Criteria:

1. People who have a history of non research related liver diseases or other diseases known to affect blood metabolism (except for controlled type II diabetes);
2. Have a history of other malignant tumors, except for fully treated basal cell carcinoma or squamous cell carcinoma and cervical carcinoma in situ;
3. Diseases requiring long-term use of immunosuppressive drugs (including steroids), including but not limited to congenital or acquired immunodeficiency diseases or active central nervous system metastatic cancer, active infection or uncontrolled heart disease;
4. Suffer from other uncontrolled serious diseases at the same time, such as unstable heart disease requiring treatment, diabetes with unsatisfactory control (fasting blood glucose>1.5 × Upper limit of normal value), mental illness and severe allergic history.
5. BMI is less than 18 or more than 25. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who met the diagnosis and criteria and were admitted to Nanfang Hospital of Southern Medical University.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Achieve the expected number of enrolled cases | 3 years
  Achieve the expected number of enrolled cases

CONTACTS AND LOCATIONS:
Overall Officials: jian guan, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No